CLINICAL TRIAL: NCT04536155
Title: Observational Study of the Quality of Life for the Chronic Pain Patients Included in a Therapeutic Education Program Focused on Relaxation Techniques
Acronym: QOLPain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Responsible Party: Sponsor
Other Study IDs: CHMS19002
Record Dates: First submitted 2020-01-07; First posted 2020-09-02 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Chronic Pain
Keywords: visualization; abdominal respiration; synchronized breathing; Sophronisation; relaxation therapy; Do In self-massage; sophrology; breathing exercise; therapeutic education
MeSH Terms: conditions — Chronic Pain | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with chronic pain
  Interventions: Other: questionnary SF36; Other: Hospital Anxiety and Depression Scale; Other: Chronic Pain Acceptance Questionnaire; Other: digital pain scale

INTERVENTIONS:
Other: questionnary SF36 — This is a validate questionnary:
  Ware et al,1992, McHorney et al, 1993, McHorney et al, 1994 French version : Author : Alain Leplège; et coll. En 2001
  Other Names: 36 items Medical Outcome Study Short Form health survey
Other: Hospital Anxiety and Depression Scale — this is a validate scale: author: Zigmond A.S., Snaith R.P. in 1983
  Other Names: HADS
Other: Chronic Pain Acceptance Questionnaire — This is a validate questionnaire:
  Fish, R., McGuire, B.E., Hogan, M., Stewart, I. & Morrison, T. (2010).
  Other Names: CPAQ
Other: digital pain scale — this is a validate scale A.N.A.E.S. February 1999

SUMMARY:
The benefit of learning psychocorporal techniques in Therapeutic Education on the quality of life of patients with chronic pain will be studied.

The purpose of this nursing research protocol is to highlight the improvement of the quality of life of chronic pain patients through psycho-physical techniques performed during group therapeutic education workshops.

DETAILED DESCRIPTION:
The study will be performed at Centre for the Study and Treatment of Pain. The patients with chronic pain will participate to a group programm of therapeutic education.

The programm consists of 9 workshops about psycho-corporal techniques performed in group.

The patients will complete questionnaries before beginning the program, at the end of the programm, 6 months after the end of the program, and 12 months after the end of program.

The questionnaries will be SF36, HADS, CPAQ, and digital pain scale.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain since more the 3months
* Patients for whom a group "relaxation techniques" program is planned and accepted by the patient

Exclusion Criteria:

* Patient with progressive cancer pain
* severe psychiatric pathology (example: psychosis, deep melancholy)
* Patient not compliant or refusing to participate in research
* Person who does not understand French, or illiterate
* Person physically unable to complete questionnaires (visually impaired or blind)
* Person protected by sections L1121-5 to L1121-8.1 of the French Public Health Code

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient with chronic pain for whom a group "relaxation techniques" programm is planned and accepted by the patient.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-10-02 (Estimated); Study Completion 2023-10-02 (Estimated)

PRIMARY OUTCOMES:
change of quality of life during the program | score at the end of the workshop compared to the score at the beginning
  SF36 score

SECONDARY OUTCOMES:
Change in quality of life | Comparison between the beginning of the program and twelve months after the end of the program.
  assessed by sf36 score
Change in anxiety and depression | Comparison at different moments in time - beginning, end, 6 months after, 12 months after
  assessed by HADS
Change in perceived pain | Assessment at the beginning of the program and 12 months after the end using a numerical pain scale
  assessed by numeric pain scale
Evolution in patient's acceptance of chronic pain:after the end | Comparison at different moments in time - beginning, end, 6 months after, 12 months after
  assessed by Chronic Pain Acceptance Questionnaire
Change in physical activity | Change in physical activity between the beginning of the program and 12 months after the end
  assessed by SF36 Physical Activity Sub-Scale

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Roullot-Pradel, Principal Investigator — CH Metropole Savoie
Locations (1):
- CH Metropole Savoie, Chambéry, France

IPD SHARING:
Plan to Share IPD: No